CLINICAL TRIAL: NCT02542982
Title: Effects of Anodal tDCS and Motor Training on Chronic Motor Deficit After Stroke
Brief Title: tDCS and Motor Training and Motor Deficit After Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Military Medical Academy, Belgrade, Serbia (Other)
Collaborators: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Tihomir Ilic, Principal Investigator, Military Medical Academy, Belgrade, Serbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFVMA/12/13-15
Record Dates: First submitted 2015-03-21; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Stroke
Keywords: tDCS; motor recovery
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment (Experimental): Group of patients on active treatment will receive intensive motor training for 45 min/day, 5 days/week, for 2 weeks, which would be preceded by 20 minutes of 2 mA anodal tDCS over the ipsilesional motor cortex.
  Interventions: Device: tDCS (Endomed 482; Enraf-Nonius B.V.)
- Sham comparator (Sham Comparator): Group of patients on sham treatment will receive intensive motor training for 45 min/day, 5 days/week, for 2 weeks, which would be preceded by sham tDCS over the ipsilesional motor cortex.
  Interventions: Device: tDCS (Endomed 482; Enraf-Nonius B.V.)

INTERVENTIONS:
Device: tDCS (Endomed 482; Enraf-Nonius B.V.) — non-invasive brain stimulation with pair of electrodes with saline-soaked pads through which the direct current of intensity of 2 mA is delivered

SUMMARY:
This study investigated the combined effects of anodal tDCS and intensive motor training (MT) vs. sham stimulation with MT (control intervention) on grip strength, motor performance and functional use of the affected arm in population of chronic stroke patients.

DETAILED DESCRIPTION:
A growing body of evidence are available regarding the effectiveness of anodal transcranial direct current stimulation (tDCS) in patients with chronic hand motor impairment as a stroke consequence.

This study investigated the combined effects of anodal tDCS and intensive motor training (MT) vs. sham stimulation with MT (control intervention) on objective evaluation of fine and gross motor hand function using simulated activities of daily living (Jebsen-Taylor hand function test), grip strength, motor performance and functional use of the affected arm in this population of patients.

Patients with chronic hand motor deficits after stroke (> 12 months) are randomly assigned to active stimulation or a control intervention arm in a double-blinded, sham-controlled, parallel design. Each group received intensive MT for 45 min/day, 5 days/week, for 2 weeks, which was preceded by 20 minutes of 2 milliampere of anodal tDCS over the ipsilesional M1 vs. sham tDCS.

Outcome measures are tested at baseline (T0), and after the intervention Day 1 (T1), after stimulation protocol completion Day 10 (T2) and 30 days later (T3).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke made by clinical features and documented by neuroimaging studies (CT or MRI scans
* stroke duration > 12 months
* severe hand deficit at stroke onset (Medical Research Council grade <2) and
* subsequently recovered to the level moderate hand deficit with presence of hand movements evaluated by the Fugl-Meyer upper-extremity Assessment (FMA) of Motor Recovery after Stroke between 28-50 points (max. 66 pts),
* spasticity between 0-2 assessed on the Modified Ashworth Scale

Exclusion Criteria:

* any clinically significant or unstable medical disorder,
* diagnosis od major depression,
* diagnosis odf substance or alcohol abuse or any neurological disorder other than stroke, including neglect, aphasia, hemianopsia and serious cognitive impairment (Mini-Mental State Examination < 24).
* any contraindications to tDCS, including histories of seizure, cerebral aneurysm, and prior surgery involving metallic implants

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Jebsen Taylor Test of Hand Function | one day, two weeks and one month
  changes of baseline summed times to complete six individual tasks (from JTT-2 to JTT7) and is performed with each hand separately

SECONDARY OUTCOMES:
hand grip force | two weeks and one month
  changes of baseline maximum grip force of the hand measured by whole-hand dynamometer
upper limb Fugl-Meyer assessment of Motor Recovery after Stroke | one day, two weeks and one month
  changes of initial score from domain of motor functions for upper limb

CONTACTS AND LOCATIONS:
Overall Officials: Tihomir V Ilic, MD, PhD, Principal Investigator — Military Medical Academy, Serbia
Locations (1):
- Clinic of Neurology, Military Medical Academy, Belgrade, Belgrade, Serbia